CLINICAL TRIAL: NCT05004870
Title: Home Examinations Researching and Understanding Submucosal Evaluations: Prospective, Virtual Study to Demonstrate Sensitivity of Submucosal Fibroids on At-home Ultrasound (Follow up to SELF-HELP Study)
Brief Title: Home Examinations Researching and Understanding Submucosal Evaluations
Acronym: HER-USE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study objective embedded into future study
Sponsor: Turtle Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 010
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Fertility Issues
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Women with a known history of submucosal fibroids (that have not been surgically removed) (Experimental)
  Interventions: Device: Transvaginal ultrasound performed by a woman herself (with HCP supervision via telemedicine)

INTERVENTIONS:
Device: Transvaginal ultrasound performed by a woman herself (with HCP supervision via telemedicine) — The ultrasound device used is cleared for HCP-supervised use in environments where healthcare is provided by trained HCPs. No changes to the design or manufacture have been made for this study.

SUMMARY:
To demonstrate that imaging via home ultrasound can identify submucosal fibroids. The image quality and submucosal fibroid detection specificity of the home imaging has already been demonstrated; the aim of this study is to generate further data for sensitivity. This will be a single visit study, with participants scanning themselves at home with healthcare professional (HCP) supervision. Targeted population is women with previously diagnosed submucosal fibroids that have not been removed. The study will be single-blinded to the image raters.

ELIGIBILITY:
Inclusion Criteria:

* Women with one or more submucosal fibroid, with appropriate attestation (see more detail below)
* Women between the ages of 18 and 49 inclusive (women 38 and younger can also receive their antral follicle count, or AFC; 39 and older will participate in uterine scanning only)
* Women with BMI up to 40
* Women located in states where the PI or sub-PI licensure is valid
* Women able to freely give consent electronically, given COVID. For the purposes of this study, this is defined as women who speak native or fluent English; and have a high school degree or equivalent, and who are otherwise, in the professional judgement of the PI, able to give informed consent

Exclusion Criteria:

* Women with expert ultrasound experience, e.g., ultrasound technologists, radiologists, OB/GYNs, Reproductive Endocrinologists
* Women with BMI over 40
* Women who do not speak English natively or fluently
* Women who have recently given birth, and have had fewer than 3 postpartum menstrual cycles
* Women who have recently had a stillbirth or abortion more than 20 weeks (subject to the 3 postpartum menstrual cycles above). Miscarriages or abortions less than 20 weeks are subject to two wait cycles
* Women who are currently pregnant or may be pregnant
* Any woman the PI believes is not capable of giving independent, informed consent
* Turtle Health employees

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-16 (Estimated); Primary Completion 2021-12-17 (Estimated); Study Completion 2021-12-17 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the at-home ultrasound for submucosal fibroids | Up to 20 minutes
  Qualified independent raters will be asked if they see a submucosal fibroid on the uterine videos. Answer options are: Yes, definitely; Almost certain; Possibly; Unlikely; No; N/A. In order to consider a fibroid present, either (1) two raters must answer "Almost certain" to having seen a submucosal fibroid or (2) one must answer "Yes definitely" to having seen a submucosal fibroid

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual metasite, Boston, Massachusetts, United States